CLINICAL TRIAL: NCT07006558
Title: Kinetic Study Of Supplementation With The Enzyme Diamine Oxidase In Patients With Histamine Intolerance
Acronym: HCB/2023/0345
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AB Biotek (Industry)
Collaborators: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: HCB/2023/0345
Record Dates: First submitted 2025-05-19; First posted 2025-06-05 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Histamine Intolerance
Keywords: diamine oxidase; histamine intolerance; safety; tolerability; pea sprout; diamine oxidase supplementation

STUDY DESIGN:
Intervention Model Description: After signing the informed consent, participants start taking the standard dose of 4.2 mg of adiDAO®Veg three times a day for a period of 2 weeks (phase 1). If the measured DAO enzyme activity levels remain unnormalized, supplementation is continued for a further 2 weeks doubling the dose (8.4 mg) (phase 2), and repeating the process of doubling doses (16.8 mg) (phase 3), 33.6 mg (phase 4), and 67.2 mg (phase 5).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Phase 1 (4.2 mg adiDAO®Veg) (Experimental): Patients receive the standard dose of 4.2 mg of adiDAO®Veg three times a day for a period of 2 weeks.
  Interventions: Dietary Supplement: Diamino Oxidase
- Phase 2 (8.4 mg adiDAO®Veg) (Experimental): If, after phase 1, the measured DAO enzyme activity levels remain unnormalized, supplementation is continued for a further 2 weeks doubling the dose to 8.4 mg of adiDAO®Veg three times a day.
  Interventions: Dietary Supplement: Diamino Oxidase
- Phase 3 (16.8 mg adiDAO®Veg) (Experimental): If, after phase 2, the measured DAO enzyme activity levels remain unnormalized, supplementation is continued for a further 2 weeks doubling the dose to 16.8 mg of adiDAO®Veg three times a day.
  Interventions: Dietary Supplement: Diamino Oxidase
- Phase 4 (33.6 mg adiDAO®Veg) (Experimental): If, after phase 3, the measured DAO enzyme activity levels remain unnormalized, supplementation is continued for a further 2 weeks doubling the dose to 33.6 mg of adiDAO®Veg three times a day.
  Interventions: Dietary Supplement: Diamino Oxidase
- Phase 5 (67.2 mg adiDAO®Veg) (Experimental): If, after phase 4, the measured DAO enzyme activity levels remain unnormalized, supplementation is continued for a further 2 weeks doubling the dose to 67.2 mg of adiDAO®Veg three times a day.
  Interventions: Dietary Supplement: Diamino Oxidase

INTERVENTIONS:
Dietary Supplement: Diamino Oxidase — The investigational product is a dehydrated power of DAO enzyme from green pea (Pisum sativum L.) sprouts (adiDAO®Veg, DR Healthcare, S.L.U., Barcelona, Spain), with an enzymatic activity > 298 mU/g (> 14,500 kHDU/g).

SUMMARY:
The present study was conducted to assess the safety and tolerability of five ascending doses of plant-based DAO enzyme supplement in subjects with symptoms of histamine intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Recent history of 2 or more symptoms associated to histamine intolerance.
* Altered activity of plasmatic DAO enzyme and/or at least one genetic variants linked to DAO deficiency (rs10156191, rs1049742, rs1049793, rs2052129).
* Not having started a dietary intervention (low histamine diet or DAO supplementation) before the start of this study.

Exclusion Criteria:

* Treatment with low-histamine diet and/or dietary DAO enzyme supplementation prior to the study.
* Pharmacological treatment with antibiotics or probiotic supplements within the last month prior to enrollment.
* Breast-feeding or pregnant women.
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events (AEs) | At "day 14", "day 28", "day 42", "day 56" and "day 70".
  Number of participants with treatment-related adverse events (AEs) experienced during the supplementation, assessed through a questionnaire.
Type of adverse effects (AEs) | At "day 14", "day 28", "day 42", "day 56" and "day 70".
  Symptoms of adverse effects (AEs) experienced during the supplementation, assessed through a questionnaire including the different body systems: gastrointestinal, CNS, respiratory, dermatological).
DAO enzymatic activity in serum using a radioextraction immunoassay | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  DAO enzymatic activity in serum (mU/mL) using a radioextraction immunoassay (REA-3H, Laboratorio Echevarne, Barcelona, Spain).

SECONDARY OUTCOMES:
Dietary habits | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Dietary habits assessed through a dietary weekly record
Histamine in 24h urine | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Histamine in 24h urine
Hemogram | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Hemogram
Glycemia | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Glycemia for safety assessment
HbA1c | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  HbA1c for safety assessment
Ionogram | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Ionogram for safety assessment
Lipid profile | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Lipid profile
C-reactive protein | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  C-reactive protein for safety assessment
Interleukin-6 | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Interleukin-6 for safety assessment
Proteinuria | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Proteinuria from urine sample
Urine sediment | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Urine sediment from urine sample for safety assessment
Gastrointestinal symptoms through Rome IV criteria | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Self-reported Gastrointestinal symptoms: Rome IV criteria
Gastrointestinal symptoms through Bristol Stool Scale | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Self-reported Gastrointestinal symptoms: Bristol Stool Scale. Score goes from Type 1 to Type 7. Higher and lower scores mean worse outcome. Middle scores (Type 3-4) are considered normal/healthy stool consistency.
Gastrointestinal symptoms through Gastrointestinal Quality of Life Index (GIQLI) | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Self-reported Gastrointestinal symptoms: Gastrointestinal Quality of Life Index (GIQLI). Score goes from 0 to 144. Higher scores indicate a better outcome.
Headaches symptoms through MIDAS questionnaire | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Self-reported Headaches symptoms through Migraine Disability Assessment Questionnaire (MIDAS) questionnaire. Score goes from 0 to >21 points. Higher scores indicate a worse outcome.
Headaches symptoms through HIT-6 questionnaire | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Self-reported Headaches symptoms through Headache Impact Test-6 (HIT-6) questionnaire. Score goes from 36 to 78. Higher scores indicate a worse outcome.
Respiratory symptoms through SNOT-22 questionnaire | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Self-reported respiratory symptoms through Sino-Nasal Outcome Test-22 (SNOT-22) questionnaire. Score goes from 0 to 110. Higher scores indicate a worse outcome.
Respiratory symptoms through Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ). Score goes from 0 to 6. Higher scores indicate a worse outcome. | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Self-reported respiratory symptoms through Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ)
Dermatological symptoms through SCORAD index | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Self-reported dermatological symptoms through SCORing Atopic Dermatitis (SCORAD) index. Score goes from 0 to 103. Higher scores indicate a worse outcome.
Dermatological symptoms through Itch Severity Scale (ISS) | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Self-reported dermatological symptoms through Itch Severity Scale. Score goes from 0 to 21. Higher scores indicate a worse outcome
Dermatological symptoms through Dermatology Life Quality Index (DLQI) | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Self-reported dermatological symptoms through Dermatology Life Quality Index (DLQI). Score goes from 0 to 20. Higher scores indicate worse outcomes.
Short-Form Health Survey (SF-36) | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Self-reported Short-Form Health Survey (SF-36) Quality of Life. Score goes from 0 to 100. Higher scores indicate a better outcome.
Creatinine (mg/dL) | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Creatinine (mg/dL) to assess renal function
Glomerular filtration rate (mL/min/1.73m2) | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Glomerular filtration rate (mL/min/1.73m2) to assess renal function
Uric acid (mg/dL) | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Uric acid (mg/dL) to assess renal function
Albuminuria (mg/L) | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Albuminuria (mg/L) to assess renal function
Albumin/creatinine ratio | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Albumin (mg/L)/creatinine (mg/dL) ratio; to assess renal function
Urine (mg/g) | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Urine (mg/g) ratio; to assess renal function
Urinary pH | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Urinary pH to assess renal function
Urine specific gravity (g/mL) | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Urine specific gravity (g/mL) to assess renal function
Aspartate Aminotransferase, ASAT (U/L) | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Aspartate Aminotransferase, ASAT (U/L) to assess hepatic function
Alanine Aminotransferase, ALAT (U/L) | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Alanine Aminotransferase, ALAT (U/L) to assess hepatic function
Gamma-Glutamyl Transferase, GGT (U/L) | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Gamma-Glutamyl Transferase, GGT (U/L) to assess hepatic function
Total Bilirubin (mg/dL) | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Total Bilirubin (mg/dL) to assess hepatic function
Alkaline Phosphatase (U/L) | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Alkaline Phosphatase (U/L) to assess hepatic function
Lactate Dehydrogenase (U/L) | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Lactate Dehydrogenase (U/L) to assess hepatic function
Total Proteins (g/L) | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Total Proteins (g/L) to assess hepatic function
Albumin (g/L) | At "baseline or day 1", "day 14", "day 28", "day 42", "day 56" and "day 70".
  Albumin (g/L) to assess hepatic function

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Serum DAO activity, participant-reported adverse effects (AEs).